CLINICAL TRIAL: NCT04497038
Title: Phase 1/2 Trial to Evaluate Cabozantinib in Patients With Advanced Hepatocellular Carcinoma With Child Pugh Class B Cirrhosis After First-Line Therapy
Brief Title: Cabozantinib in Patients With Advanced Hepatocellular Carcinoma With Child Pugh Class B Cirrhosis After First-Line Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: loss of funding
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2020.007; HUM00176488 (Other: University of Michigan)
Record Dates: First submitted 2020-06-29; First posted 2020-08-04 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
MeSH Terms: interventions — cabozantinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cabozantinib (Experimental): Cabozantinib 20-60 mg by mouth once daily.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Patients will receive therapy with cabozantinib. Dosage in the trial will start at 40 mg PO daily. Each patient will be assessed for the development of toxicity according to the NCI Common Terminology Criteria for Adverse Events, version 5.0. Dose adjustments may be made per the Time-To-Event modification of the Continual Reassessment Method (TITE-CRM). The maximum dosage will be 60 mg PO daily and the minimum will be 20 mg PO daily.

SUMMARY:
The aim of this study is to determine the safety and efficacy of cabozantinib in the management of unresectable or metastatic hepatocellular carcinoma (HCC) with underlying Child-Pugh class B cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a radiologically consistent (early enhancement and delayed enhancement washout) or pathologically confirmed diagnosis of hepatocellular carcinoma that is not eligible for curative resection, transplantation, or ablative therapies.
* Prior radiation, liver directed therapy (including bland, chemo- or radioembolization, or ablation), or hepatic resection are permitted if ≥4 weeks from start of therapy. Extra-hepatic palliative radiation is permitted if completed ≥2 weeks prior to first dose of study therapy and the patient has recovered to ≤ grade 1 toxicity.
* Patients must have radiographically measurable disease (RECIST1.1) in at least one site not previously treated or with progression after radiation or liver directed therapy (including bland, chemo- or radio-embolization, or ablation) either within the liver or in a metastatic site.
* Patients must have either progressed or deemed intolerant of first-line systemic therapy. More than one line of systemic therapy is not permitted. The last dose should be at least 2 weeks from first dose of study therapy. Prior treatment may not contain cabozantinib.
* Recovery to ≤ grade 1 from toxicities related to any prior treatments, unless the AEs were clinically non-significant and/or stable on supportive therapy
* Must have a Child-Pugh score of B7 or B8
* Must have an ECOG performance status of 0-1.
* Ability to understand and willingness to sign IRB-approved informed consent.
* Willing to provide archived tissue, if available, from a previous diagnostic biopsy.
* Must be able to tolerate CT and/or MRI with contrast.
* Adequate organ function obtained ≤ 2 weeks prior to enrollment.

Exclusion Criteria:

* Must not have uncontrolled ascites (requiring paracentesis within 3 months of screening) or hepatic encephalopathy requiring hospitalization (within 6 months of screening)
* Must not have prior history of organ transplantation.
* No known brain metastasis unless adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before registration. Eligible subjects must have been without corticosteroid treatment at the time of registration.
* Must not have undergone a major surgery (e.g., GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (e.g., simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications from prior surgery are not eligible.
* Must not have an active second malignancy other than non-melanoma skin cancer or cervical carcinoma in situ. Patients with history of malignancy are eligible provided primary treatment of that cancer was completed > 1 year prior to enrollment and the patient is free of clinical or radiologic evidence of recurrent or progressive malignancy.
* Must not have uncontrolled, significant intercurrent or recent illness including, but not limited to the following conditions:

  * Cardiovascular disorders (Congestive heart failure or uncontrolled hypertension; or stroke, myocardial infarction, or other ischemic or thromboembolic event within 6 months before first dose)
  * Gastrointestinal disorders, including those associated with a high risk of perforation or fistula formation
  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon of red blood or other history of significant bleeding within 12 weeks before first dose
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation
  * Lesions invading or encasing any major blood vessels except thromboses of portal/hepatic vasculature attributed to underlying liver disease and/or liver tumor
  * Other clinically significant disorders that would preclude safe study participation (serious non-healing wound/ulcer/bone fracture; uncompensated/symptomatic hypothyroidism; known HIV)
* Must not have untreated or incompletely treated varices with bleeding or high risk for bleeding. Subjects treated with adequate endoscopic therapy (in accordance with institutional standards) without any episodes of recurrent overt GI bleeding requiring transfusion or hospitalization for at least 6 months prior to study entry are eligible
* Must not have a psychiatric illness, other significant medical illness, or social situation (such as involuntary incarceration) which, in the investigator's opinion, would limit compliance or ability to comply with study requirements
* Women must not be pregnant or breastfeeding since cabozantinib may harm the fetus or child.
* Women of child-bearing potential (not surgically sterilized and between menarche and 1-year post menopause) and men must agree to use 2 methods of adequate contraception (hormonal plus barrier or 2 barrier forms) OR abstinence prior to study entry, for the duration of study participation, and for 4 months following completion of study therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Prisoners or subjects who are involuntarily incarcerated, or compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness would be excluded.
* Concomitant treatment with strong inducers or inhibitors of CYP3A4 is not allowed. Patients must discontinue the drug(s) at least 14 days prior to first study dose on the study.
* Concomitant anticoagulation with oral anticoagulants (e.g. warfarin, direct thrombin and factor Xa inhibitors), or platelet inhibitors (e.g. clopidogrel) is not allowed.
* Must not have corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaibhav Sahai, MBBS, MS, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabozantinib: Cabozantinib 20-60 mg by mouth once daily.
  Patients received therapy with cabozantinib. Dosage in the trial will start at 40 mg PO daily. Each patient will be assessed for the development of toxicity according to the NCI Common Terminology Criteria for Adverse Events, version 5.0. Dose adjustments may be made per the Time-To-Event modification of the Continual Reassessment Method (TITE-CRM). The maximum dosage will be 60 mg PO daily and the minimum will be 20 mg PO daily.
Period: Overall Study
Arm/Group | Cabozantinib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of DLT Events to Occur
Description: MTD/RP2D determined by dose limiting toxicities (DLT) during the first 29 days of therapy. DLTs are outlined in the protocol and assessed per the NCI CTCAE v5.0. The MTD/RP2D will be determined as the dose level with the highest probability of DLT not exceeding 35%.
Time Frame: Up to 29 days after initiating treatment
Measure: Number; unit: Number of DLT events to occur
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
Number of DLT events to occur | 0

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS defined as time from date of treatment to date of radiological or clinical progressing (leading to withdrawal from the study), or death from any cause, whichever comes first. PFS will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: 1.7 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
Months | 5.42 [4.30 to 5.51]

3. Secondary Outcome: Median Time to Progression (TTP)
Description: TTP defined as time from date of treatment to date of radiological or clinical progression (leading to withdrawal from the study).
Time Frame: 1.7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
months | 5.42 [4.30 to 5.51]

4. Secondary Outcome: Overall Survival (OS)
Description: Patients will be followed for up to 2 years from treatment discontinuation or until death, whichever comes first, or 3 years after first date of treatment initiation for those that remain on treatment. OS will be estimated using the product-limit method of Kaplan and Meier.
Time Frame: 1.7 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
months | 9.33 [7.91 to 13.40]

5. Secondary Outcome: Overall Response Rate (ORR) (Partial Response + Complete Response)
Description: ORR (PR + CR) per RECIST v1.1 criteria during active study treatment.
Time Frame: 1.7 years
Measure: Number; unit: participants with a PR or CR
Arm/Group | Cabozantinib
Number analyzed (Participants) | 3
participants with a PR or CR | 0

6. Secondary Outcome: Pharmacokinetic (PK) Profile: Elimination Clearance (L/hr)
Description: Blood draws pre-dose, every 2 weeks until the start of cycle 3
Time Frame: Up to 2 months
Population: PK data was never conducted as study was halted prematurely
Arm/Group | Cabozantinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1.7 years
Groups:
- Cabozantinib: Cabozantinib 20-60 mg by mouth once daily.
  Patients received therapy with cabozantinib. Dosage in the trial will start at 40 mg PO daily. Each patient will be assessed for the development of toxicity according to the NCI Common Terminology Criteria for Adverse Events, version 5.0. Dose adjustments may be made per the Time-To-Event modification of the Continual Reassessment Method (TITE-CRM). The maximum dosage will be 60 mg PO daily and the minimum will be 20 mg PO daily.
  Due to low number of enrolled patients, we cannot separate based on dose level in order to maintain confidentiality.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=3)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (3)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=3)
Hypothyroidism (Endocrine disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
burn (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04497038/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT04497038/ICF_001.pdf